CLINICAL TRIAL: NCT06381050
Title: An Open-label, Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-7631 for Injection in Patients With Advanced Solid Tumors
Brief Title: The Clinical Study of SHR-7631 for Injection in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-7631-101
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-7631 (Experimental)
  Interventions: Drug: SHR-7631

INTERVENTIONS:
Drug: SHR-7631 — The total dosage of SHR-7631 was calculated according to the weight weighing results of the subjects before each administration, and was administered by intravenous drip.

SUMMARY:
This study is an open-label, phase I clinical trial of SHR-7631 in patients with advanced solid tumors. The whole study is divided into three stages: dose escalation, dose expansion and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment, or standard treatment is not applicable currently;
2. Have at least one measurable tumor lesion per RECIST v1.1 (subject with only non-target tumor lesion will be permitted if he/she is planned to participant in dose escalation stage or with mCRPC);
3. ECOG performance status of 0-1;
4. Life expectancy ≥ 12 weeks;
5. Adequate bone marrow and organ function
6. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
7. Age 18 to 75 years old (including both ends), gender is not limited;

Exclusion Criteria:

1. Patients with active central nervous system metastases or meningeal metastases;
2. Ongoing or previous anti-tumor therapies within 4 weeks prior to the first dose of study drug;
3. Prior treatment with antibody-drug conjugate (ADC) consisting of topoisomerase I inhibitors;
4. History of serious cardiovascular and cerebrovascular diseases;
5. Severe infection within 4 weeks prior to the first dose;
6. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum administered dose (MAD) | 12 months
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) (CTCAE v5.0) | 36 months

SECONDARY OUTCOMES:
PK parameter: Tmax | 36 months
PK parameter: Cmax | 36 months
PK parameter: AUC0-t | 36 months
PK parameter: AUC0-∞ | 36 months
PK parameter: t1/2 | 36 months
PK parameter: MRT (mean residence time) | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangzhou

IPD SHARING:
Plan to Share IPD: Undecided